CLINICAL TRIAL: NCT01715948
Title: A Comparison Between Wireless CROS and Bone-anchored Hearing Devices for Single-Sided Deafness: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manohar Bance (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Sponsor-Investigator, Manohar Bance, Staff Physician Division of Otolaryngology, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDHA-RS/2013-118
Record Dates: First submitted 2012-10-23; First posted 2012-10-29 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Unilateral Hearing Loss; Unilateral Deafness
Keywords: CROS hearing aid; Bone-anchored hearing device
MeSH Terms: conditions — Hearing Loss, Unilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CROS hearing aid (Experimental): The CROS uses two hearing aids that fit behind each ear. The hearing aid fitted with a retainer earhook on the side of the poor ear houses a microphone and a transmitter. The hearing aid fitted on the normal ear side houses a receiver that is connected to a slim tube and open ear tip. The CROS does not amplify sound but rather transmits sound from the side of the unaidable ear to the contralateral ear, overcoming the head shadow effect that presents with SSD.
  Interventions: Device: CROS hearing aid
- Bone-anchored hearing device (BAHD) (Experimental): The BAHD (such as the Baha by Cochlear or Bone-Bridge by MED-EL) also helps to alleviate the negative effect of head shadow and the difficulty with speech perception in noise that present with SSD. Also known as an osseointegrated aural prosthesis, the BAHD is implanted in individuals with SSD to stimulate the ear with the normal cochlea. The BAHD requires that a titanium screw be surgically implanted in the temporal bone on the side of the poor ear. This titanium screw is connected to a percutaneous abutment. An electromechanical sound processor (external transducer) is coupled onto the abutment and can be removed when necessary. Sound can now be routed to the better ear by transcranial bone conduction.
  Interventions: Device: Bone-anchored hearing device (BAHD)

INTERVENTIONS:
Device: CROS hearing aid — Participants were randomly assigned to be fitted with the CROS hearing aid either at the end of the first visit or at the end of the second visit. They were given a 2-week trial with the CROS and asked to refrain from wearing their BAHD during that time. At the end of the first visit, four participants were fitted with the CROS hearing aid and were subsequently tested with this device on their second visit, at which time they were instructed to use the BAHD for the next 2 weeks. This protocol was reversed in the other four participants, with testing after each device experience. Both devices were compared on head shadow effect reduction, speech perception measures in quiet and in noise, self-assessment questionnaires, and daily diaries.
  Other Names: Unitron Tandem 4 CROS hearing aid
  Arms: CROS hearing aid
Device: Bone-anchored hearing device (BAHD) — All participants had received BAHD implantation prior to the study. They were randomly selected to continue wearing their BAHD for 2 weeks following the end of the first visit or the end of the second visit. Both devices were compared on head shadow effect reduction, speech perception measures in quiet and in noise, self-assessment questionnaires, and daily diaries.
  Arms: Bone-anchored hearing device (BAHD)

SUMMARY:
People with single-sided deafness (SSD) have significant hearing loss in one ear and normal or near normal hearing in the other ear. Those living with SSD experience several communication difficulties, particularly when listening to speech in the presence of background noise. This problem is worse in situations where the noise is on the side of the good ear and the speech is on the side of the poor ear.

The Bone-anchored hearing device (BAHD) and the Contralateral Routing of Signals (CROS) hearing aid are two intervention methods designed to improve hearing in people who have significant hearing loss in one ear only. The BAHD is a surgically implanted device which also includes an external processor; sounds from the poor ear are transmitted to the good ear through skull vibrations. The CROS does not involve surgery; instead a hearing aid is fitted behind each ear, and the sounds on the side of the poor ear are wirelessly transmitted to the good ear.

The majority of previous studies comparing the BAHD to the CROS have used older CROS models with basic technology and a wire along the neck to send sounds from the poor ear to the good ear. There is a lack of studies comparing newer digital wireless CROS hearing aids to the BAHD. The current research will compare the effect of the BAHD and CROS hearing aid on speech perception scores when listening to speech in quiet and in noise. The research will also investigate participants' reported benefits with each device during everyday situations. In order to compare the BAHD and CROS, individuals who already have been implanted with a BAHD will be given a trial period with a new wireless digital CROS hearing aid.

The research hypothesis states that the CROS hearing aid will be as equally beneficial or greater than the BAHD in improving hearing and participant benefit. If the findings support the hypothesis that the CROS offers just as much benefits as the BAHD, or is an even better alternative, more individuals with SSD may choose to avoid surgery and decide to receive a CROS hearing aid instead.

DETAILED DESCRIPTION:
Users of the BAHD will be given a 2-week trial period with the Unitron Tandem CROS hearing aid. Participants will be randomly assigned to wear either their BAHD for two weeks or the trial CROS for two weeks. There will be a total of three visits made to the clinic.

During each visit:

* Participants' hearing will be tested (either with the BAHD, the CROS, or without wearing any device).
* Speech perception ability will be tested in quiet and in noise conditions (either while wearing the BAHD, the CROS, or no device).
* Participants will be asked to complete two standardized questionnaires on the perceived benefits that the BAHD or the CROS provides.

In addition, participants will be asked to fill out a short diary form every day, for a two-week period, to report the situations in which they wore the device.

ELIGIBILITY:
Inclusion Criteria:

* Adults with unilateral deafness (hearing loss in only one ear) who received BAHD surgery less than 3 years ago
* Severe to profound hearing loss in the poor ear and normal hearing in the good ear
* English speaking

Exclusion Criteria:

* Adults who underwent BAHD surgery more than 3 years ago
* Adults with hearing loss in both ears
* Adults who received a BAHD to treat a condition other than unilateral deafness (such as bilateral conductive hearing loss)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manohar Bance, FRCS, Principal Investigator — Capital Health, Canada; Rachel Caissie, Ph.D., Principal Investigator — Dalhousie University; Jennifer Finbow, B.Sc., Principal Investigator — Dalhousie University

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Contralateral Routing of Signals (CROS) Hearing Aid: Participants who have been implanted with a bone-anchored hearing device (BAHD) over the past three years will be given a two-week trial period with a Contralateral Routing of Signals (CROS) hearing aid. The CROS uses two hearing aids that fit behind each ear. The hearing aid fitted on the side of the poor ear houses a microphone and a transmitter. The hearing aid fitted on the normal ear side houses a receiver that is connected to an open ear tip. Sounds on the side of the poor ear are picked up by the microphone and transmitted to the opposite normal ear, overcoming the head shadow effect that presents with unilateral deafness.
  Both devices were compared on head shadow effect reduction, speech perception measures in quiet and in noise, self-assessment questionnaires, and daily diaries.
Period: Overall Study
Arm/Group | Contralateral Routing of Signals (CROS) Hearing Aid
Started | 9
Completed | 8
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- A Comparison Between Wireless CROS and BAHD for SSD: Participants who have been implanted with a BAHD over the past three years will be given a two-week trial period with a CROS hearing aid. The CROS uses two hearing aids that fit behind each ear. The hearing aid fitted on the side of the poor ear houses a microphone and a transmitter. The hearing aid fitted on the normal ear side houses a receiver that is connected to an open ear tip. Sounds on the side of the poor ear are picked up by the microphone and transmitted to the opposite normal ear, overcoming the head shadow effect that presents with unilateral deafness.
  CROS hearing aid: BAHD users will be fitted with the CROS hearing aid for a two-week trial period. Their hearing abilities with the CROS hearing aid will be compared to their hearing abilities with their BAHD over a two-week period.
Arm/Group | A Comparison Between Wireless CROS and BAHD for SSD
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 54 [44 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Region of Enrollment [Number; unit: participants]
  Canada | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of 5 Key Words Within 6 Sentence Lists Repeated Correctly in the Presence of Multitalker Noise
Description: One speech-in-noise test (QuickSIN) presented four lists of six pre-recorded sentences at 50 dB hearing level (HL) in soundfield. Multitalker noise was presented together with the target sentence and increased at a fixed number of dB with the completion of each sentence. The multitalker noise was initially presented at 25 dB HL (signal-to-noise ratio - SNR of 25 dB), and increased by 5 dB after each sentence until the multitalker noise was of equal intensity with the final sentence (SNR of 0 dB). In one condition, two lists of sentences were presented to the participant at 0 degrees with the multitalker noise delivered at 90 degrees to the poor ear. In the other condition, two different lists of sentences were presented to the participant at 0 degrees with the multitalker noise delivered at 90 degrees to the better ear. The two scores derived from the two different lists of sentences presented within each condition were averaged. A low score indicates better performance.
Time Frame: The QuickSIN unaided was administered at baseline, an average of 2 weeks (with CROS or BAHD) and an average of 4 weeks (with opposite device not previously tested).
Measure: Mean (95% Confidence Interval); unit: words
Groups:
- QuickSIN Noise to Better Ear Unaided: Two different lists of sentences presented at 0 degree azimuth and multitalker noise presented at 90 degrees azimuth to the better ear while wearing no device. The multitalker noise increases with each sentence presentation such that the signal-to-noise ratio decreases from 25 to 0 dB, in 5-dB steps, over the six sentences.
- QuickSIN Noise to Better Ear With BAHD: Two different lists of sentences presented at 0 degree azimuth and multitalker noise presented at 90 degrees azimuth to the better ear while wearing the BAHD.
- QuickSIN Noise to Better Ear With CROS: Two different lists of sentences presented at 0 degree azimuth and multitalker noise presented at 90 degrees azimuth to the better ear while wearing the CROS.
- QuickSIN Noise to Poorer Ear Unaided: Two different lists of sentences presented at 0 degree azimuth and multitalker noise presented at 90 degrees azimuth to the poorer ear while wearing no device.
- QuickSIN Noise to Poorer Ear With BAHD: Two different lists of sentences presented at 0 degree azimuth and multitalker noise presented at 90 degrees azimuth to the poorer ear while wearing the BAHD.
- QuickSIN Noise to Poorer Ear With CROS: Two different lists of sentences presented at 0 degree azimuth and multitalker noise presented at 90 degrees azimuth to the poorer ear while wearing the CROS.
Arm/Group | QuickSIN Noise to Better Ear Unaided | QuickSIN Noise to Better Ear With BAHD | QuickSIN Noise to Better Ear With CROS | QuickSIN Noise to Poorer Ear Unaided | QuickSIN Noise to Poorer Ear With BAHD | QuickSIN Noise to Poorer Ear With CROS
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
words | 5.44 [4.461 to 6.419] | 3.5 [2.646 to 4.354] | 4.75 [3.815 to 5.685] | -1.75 [-2.346 to -1.154] | 0.75 [-0.089 to 1.589] | 2.38 [1.786 to 2.974]

2. Primary Outcome: Percentage of Words Recognized
Description: Word recognition was tested with the recorded version of the Central Institute for the Deaf (CID) W-22 (Auditec of St. Louis), with a different list of 25 monosyllabic words presented at 50 dB HL in three randomized listening conditions. In the first condition, one list was presented at 50 dB HL at 90 degrees to the poor ear in quiet. In the second condition, the words were presented at 50 dB HL at 0 degrees while multitalker noise was presented at 45 dB HL at 90 degrees to the poor ear. In the final condition, the words were presented at 50 dB HL at 0 degrees while multitalker noise was delivered at 45 dB HL at 90 degrees to the better ear.
Time Frame: Word recognition testing (unaided) occurred at baseline, an average of 2 weeks (with CROS or BAHD) and an average of 4 weeks (with opposite device not previously tested)..
Population: The researchers chose not to include a condition with words presented at 90 degrees to the better ear in quiet.
Measure: Mean (95% Confidence Interval); unit: Percentage of words perceived correctly
Groups:
- WRS Noise to Better Ear: Word recognition was tested with words presented from the front and multitalker noise (at 45 dB HL) at 90 degrees azimuth to the better ear. This occurred across three randomized listening conditions: unaided, BAHD and CROS.
- WRS Noise to Poorer Ear: Word recognition was tested with words presented from the front and multitalker noise (at 45 dB HL) at 90 degrees azimuth to the poorer ear. This occurred across three randomized listening conditions: unaided, BAHD and CROS.
- WRS in Quiet to Poorer Ear: Word recognition was tested with no noise (quiet) with words presented at 90 degrees azimuth to the poorer ear. This occurred across three randomized listening conditions: unaided, BAHD and CROS.
Arm/Group | WRS Noise to Better Ear | WRS Noise to Poorer Ear | WRS in Quiet to Poorer Ear
Number analyzed (Participants) | 8 | 8 | 8
Percentage of words perceived correctly
  Unaided Condition | 48.5 [42.23 to 54.77] | 78 [74.56 to 81.44] | 96 [94.25 to 97.75]
  BAHD Condition | 62.5 [55.81 to 69.19] | 77 [70.97 to 83.03] | 97 [94.77 to 99.23]
  CROS Condition | 62 [57.48 to 66.52] | 66.5 [60.22 to 72.78] | 94.5 [91.85 to 97.15]

3. Primary Outcome: Speech Spatial Qualities Questionnaire (SSQ)
Description: The Speech Spatial Qualities Questionnaire (SSQ) was given to assess the self-perceived benefits provided by the device that was worn the previous 2 weeks. The SSQ requires participants to rate their perceived hearing ability for 49 scenarios using a 10-point scale, ranging from 0 ("Not at all") to 10 ("Perfectly"). A score higher than 0 for each listening scenario shows some benefit of the device, while a score of 10 indicates the device was extremely beneficial. Therefore, a lower score indicated poorer self-perceived benefit from the device (representing a worse outcome), while a higher score indicated greater self-perceived benefit from the device (representing a better outcome). To obtain individual scores for the SSQ questionnaire, the ratings for each listening scenario were summed. The mean, minimum and maximum scores for each subscale of the SSQ across all participants were also determined.
Time Frame: Administered at the end of a 2 week trial with the CROS and at the end of a 2 week use of the BAHD.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- SSQ Subscale - Speech (BAHD): Participants rated the effectiveness of the BAHD for listening situations included in the Speech subscale of the SSQ on a 10-point scale.
- SSQ Subscale - Speech (CROS): Participants rated the effectiveness of the CROS for listening situations included in the Speech subscale of the SSQ on a 10-point scale.
- SSQ Subscale - Spatial (BAHD): Participants rated the effectiveness of the BAHD for listening situations included in the Spatial subscale of the SSQ on a 10-point scale.
- SSQ Subscale - Spatial (CROS): Participants rated the effectiveness of the CROS for listening situations included in the Spatial subscale of the SSQ on a 10-point scale.
- SSQ Subscale - Qualities (BAHD): Participants rated the effectiveness of the BAHD for listening situations included in the Qualities subscale of the SSQ on a 10-point scale.
- SSQ Subscale - Qualities (CROS): Participants rated the effectiveness of the CROS for listening situations included in the Qualities subscale of the SSQ on a 10-point scale.
Arm/Group | SSQ Subscale - Speech (BAHD) | SSQ Subscale - Speech (CROS) | SSQ Subscale - Spatial (BAHD) | SSQ Subscale - Spatial (CROS) | SSQ Subscale - Qualities (BAHD) | SSQ Subscale - Qualities (CROS)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
units on a scale | 5.56 [5.112 to 6.008] | 5.79 [5.365 to 6.215] | 4.24 [3.727 to 4.753] | 4.45 [3.702 to 5.198] | 6.89 [6.431 to 7.349] | 7.12 [6.43 to 7.81]

ADVERSE EVENTS:
Groups:
- BAHD: The intervention during which the BAHD was trialed as part of the cross-over design
- CROS Aid: The intervention during which the CROS aid was trialed as part of the cross-over design
Arm/Group | BAHD | CROS Aid
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/0
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
The sample size was small and included only one male. The trial period of two weeks was short and may not have provided enough time for participants to adjust to the new CROS. The long-term benefit of both hearing devices needs to be assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No